CLINICAL TRIAL: NCT03936595
Title: Investigation on the Recovery Kinetics of Performance, Muscle Damage and Neuromuscular Fatigue Indicators, Following Different Protocols for Muscle Power Development
Brief Title: Recovery of Performance, Muscle Damage and Neuromuscular Fatigue Following Muscle Power Training
Acronym: PoTrRec
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: There was a high drop-out rate and we were unable to recruit new subjects.
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Ioannis G. Fatouros, Professor, University of Thessaly
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Power Training-Recovery UTH
Record Dates: First submitted 2019-04-30; First posted 2019-05-03 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Power Training Exercise Protocols

STUDY DESIGN:
Intervention Model Description: Each participant will perform in a random order all four different experimental conditions
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Core exercises protocol (Experimental): Participants will perform 4 core exercises
  Interventions: Other: Core exercises protocol
- Structural exercises protocol (Experimental): Participants will perform 4 structural (Olympic lifting) exercises
  Interventions: Other: Structural exercises protocol
- Accentuated eccentric load exercises protocol (Experimental): Participants will perform 4 exercises with eccentric loading
  Interventions: Other: Accentuated eccentric load exercises protocol
- Control condition (Other): Participants will perform all the measurements that are comprised in the experimental conditions without performing any exercise protocol
  Interventions: Other: Control condition

INTERVENTIONS:
Other: Core exercises protocol — Participants will perform:
  1. Squats, 4 sets of 5 repetitions at 60% 1RM
  2. Deadlifts, 4 sets of 5 repetitions at 60% 1RM
  3. Lunges, 4 sets of 5 repetitions at 60% 1RM
  4. Step ups, 4 sets of 5 repetitions at 60% 1RM
  Arms: Core exercises protocol
Other: Structural exercises protocol — Participants will perform:
  1. Snatch, 4 sets of 5 repetitions at 60% 1RM
  2. Hang clean, 4 sets of 5 repetitions at 60% 1RM
  3. Push jerk, 4 sets of 5 repetitions at 60% 1RM
  4. Split push jerk, 4 sets of 5 repetitions at 60% 1RM
  Arms: Structural exercises protocol
Other: Accentuated eccentric load exercises protocol — Participants will perform:
  1. Deadlifts - squat jump, 4 sets of 5 repetitions at 30% body mass (BM)
  2. Step down - squat jump, 4 sets of 5 repetitions at 30% BM
  3. Step down - lunges, 4 sets of 5 repetitions at 30% BM
  4. Hip thrusts, 4 sets of 5 repetitions at 30% BM
  Arms: Accentuated eccentric load exercises protocol
Other: Control condition — Participants will perform all the measurements that are comprised in the experimental conditions without performing any exercise protocol
  Arms: Control condition

SUMMARY:
Muscle power is one of the most important parameters in almost every athletic action, and expresses the ability of the human muscle to produce great amounts of force with the greatest possible speed. Thus, muscle power is critical for high performance in athletic actions such as jumping, throwing, change of direction and sprinting. For enhancing their muscle power, athletes comprise several resistance training programs as part of their training. Muscle power training comprises of eccentric muscle actions, and the magnitude of these actions depend on the emphasis that is given on the concentric or eccentric action, respectively, of the muscles during the exercises. However, eccentric muscle action, especially when unaccustomed, can lead to exercise-induced muscle damage (EIMD), and deterioration of muscle performance.

Despite the fact that muscle power training comprises eccentric muscle actions, and consequently can lead to muscle injury and muscle performance reduction during the following days, the recovery kinetics after acute muscle power training have not been adequately studied. However, information regarding the recovery of the muscles after a power training protocol, is critical for the correct design of a training microcycle, and the reduction of injury risk.

The aim of the present study is to investigate the muscle injury provoked after acute muscle power training using three different power training exercise protocols. Additionally, we will examine the effect of these protocols on muscle performance and neuromuscular fatigue indices.

DETAILED DESCRIPTION:
Muscle power is one of the most important parameters in almost every athletic action, and expresses the ability of the human muscle to produce great amounts of force with the greatest possible speed. Thus, muscle power is critical for high performance in athletic actions such as jumping, throwing, change of direction and sprinting.

For enhancing their muscle power, athletes comprise several resistance training programs as part of their training. Core exercises as long as Olympic lifting has been used in muscle power training. The loads that are applied regarding the accomplishment of the most favorable power production are varying. Training load of 0% 1RM favored power production at the countermovement squat jump, while loads of 56% 1rm and 80% 1RM, favored the power production at squat and hang clean, respectively. Additionally, In the recent years, accentuated eccentric training has been proposed as a new training method for the enhancement of muscle power. This method emphasizes the eccentric component of the muscle contraction, and there is evidence supporting the greater production of muscle force after accentuated eccentric training compared with the typical resistance exercise training method.

Taking the above into consideration, muscle power training comprises of eccentric muscle actions, and the magnitude of the eccentric component depends on the emphasis that is given on the concentric or eccentric action, respectively, of the muscles during the exercises. However, eccentric muscle action, especially when unaccustomed, can lead to exercise-induced muscle damage (EIMD). Although concentric and isometric exercise may also lead to muscle injury, the amount of damage after eccentric muscle contractions is greater. EIMD, amongst others, is accompanied by increased levels of creatine kinase (CK) into the circulation, increased delayed onset of muscle soreness (DOMS), reduction of force production, reduction of flexibility speed.

Despite the fact that muscle power training comprises eccentric muscle actions, and consequently can lead to muscle injury and muscle performance reduction during the following days, the recovery kinetics after acute muscle power training protocols have not been adequately studied. However, information regarding the recovery of the muscles after a power training protocol, is critical for the correct design of a training microcycle, and the reduction of injury risk.

The aim of the present study is to investigate the muscle injury provoked after muscle acute power training using three different power training exercise protocols. Additionally, the effect of these protocols on muscle performance and neuromuscular fatigue indices will be examined.

ELIGIBILITY:
Inclusion Criteria:

* No recent history of musculoskeletal injury
* No use of ergogenic supplements and drugs
* No use of anti-inflammatory and antioxidant supplements (> 6 months)
* No participation at intense eccentric exercise for at least 3 days before protocols

Exclusion Criteria:

* Recent history of musculoskeletal injury
* Use of ergogenic supplements and drugs
* Use of anti-inflammatory and antioxidant supplements (< 6 months)
* Participation at intense eccentric exercise for at least 3 days before protocols

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2019-06-16 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Change on delayed onset of muscle soreness (DOMS), in the knee flexors (KF) and extensors (KE) of both limbs | Prior to, immediately after, 1, 2, 3 days after the end of the experimental protocol
  Participants will perform three repetitions of a full squat movement, and rate their soreness level in knee flexors and extensors on a visual analog scale from 1 to 10 (VAS, with "no pain" at one end and "extremely sore" at the other), using palpation of the belly and the distal region of relaxed knee extensors and flexors.
Change on countermovement jump (CMJ) height | Prior to, immediately after, 1, 2, 3 days after the end of the experimental protocol
  CMJ height will be measured in 3 maximal efforts (the best jump will be recorded) on an Ergojump contact platform
Change on isometric peak torque of the knee extensors (KE) | Prior to, immediately after, 1, 2, 3 days after the end of the experimental protocol
  Isometric peak torque of the KE will be measured on an isokinetic dynamometer at 60◦/sec
Change on isometric peak torque of the knee flexors (KF) | Prior to, immediately after, 1, 2, 3 days after the end of the experimental protocol
  Isometric peak torque of the KF will be measured on an isokinetic dynamometer at 60◦/sec
Change on concentric isokinetic peak torque of the knee extensors (KE) | Prior to, immediately after, 1, 2, 3 days after the end of the experimental protocol
  Concentric peak torque of the KE will be measured on an isokinetic dynamometer at 60◦/sec
Change on concentric isokinetic peak torque of the knee flexors (KF) | Prior to, immediately after, 1, 2, 3 days after the end of the experimental protocol
  Concentric peak torque of the KF will be measured on an isokinetic dynamometer at 60◦/sec
Change one eccentric isokinetic peak torque of the knee extensors (KE) | Prior to, immediately after, 1, 2, 3 days after the end of the experimental protocol
  Eccentric peak torque of the KE will be measured on an isokinetic dynamometer at 60◦/sec
Change on eccentric isokinetic peak torque of the knee flexors (KF) | Prior to, immediately after, 1, 2, 3 days after the end of the experimental protocol
  Eccentric peak torque of the KF will be measured on an isokinetic dynamometer at 60◦/sec
Change on the concentration of plasma CK activity | Prior to, immediately after, 1, 2, 3 days after the end of the experimental protocol
  Plasma CK activity will be measured with a biochemical analyzer
Change on the concentration of blood lactate | Prior to, and immediately after the end of the experimental protocol
  Lactate will be measured with a portable lactate analyzer using capillary blood

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis G Fatouros, PhD, Principal Investigator — University of Thessaly
Locations (1):
- Laboratory of Exercise Biochemistry, Exercise Physiology,and Sports Nutrition, School of Physical Education and Sport Science, University of Thessaly, Trikala, Thessaly, Greece

REFERENCES:
- [Background] Cormie P, McCaulley GO, Triplett NT, McBride JM. Optimal loading for maximal power output during lower-body resistance exercises. Med Sci Sports Exerc. 2007 Feb;39(2):340-9. doi: 10.1249/01.mss.0000246993.71599.bf. PMID 17277599
- [Background] Baird MF, Graham SM, Baker JS, Bickerstaff GF. Creatine-kinase- and exercise-related muscle damage implications for muscle performance and recovery. J Nutr Metab. 2012;2012:960363. doi: 10.1155/2012/960363. Epub 2012 Jan 11. PMID 22288008
- [Background] Deli CK, Fatouros IG, Paschalis V, Georgakouli K, Zalavras A, Avloniti A, Koutedakis Y, Jamurtas AZ. A Comparison of Exercise-Induced Muscle Damage Following Maximal Eccentric Contractions in Men and Boys. Pediatr Exerc Sci. 2017 Aug;29(3):316-325. doi: 10.1123/pes.2016-0185. Epub 2017 Feb 6. PMID 28165870
- [Background] Jamurtas AZ, Theocharis V, Tofas T, Tsiokanos A, Yfanti C, Paschalis V, Koutedakis Y, Nosaka K. Comparison between leg and arm eccentric exercises of the same relative intensity on indices of muscle damage. Eur J Appl Physiol. 2005 Oct;95(2-3):179-85. doi: 10.1007/s00421-005-1345-0. Epub 2005 Jul 9. PMID 16007451
- [Background] Kyrolainen H, Avela J, McBride JM, Koskinen S, Andersen JL, Sipila S, Takala TE, Komi PV. Effects of power training on muscle structure and neuromuscular performance. Scand J Med Sci Sports. 2005 Feb;15(1):58-64. doi: 10.1111/j.1600-0838.2004.00390.x. PMID 15679573
- [Background] Walker S, Blazevich AJ, Haff GG, Tufano JJ, Newton RU, Hakkinen K. Greater Strength Gains after Training with Accentuated Eccentric than Traditional Isoinertial Loads in Already Strength-Trained Men. Front Physiol. 2016 Apr 27;7:149. doi: 10.3389/fphys.2016.00149. eCollection 2016. PMID 27199764